CLINICAL TRIAL: NCT06524102
Title: Evaluation of the Efficacy of Annexin Columns (MACS) in Patients With Altered Sperm FISH Undergoing Assisted Reproductive Techniques
Brief Title: The Aim of This Study is to Determine the Incidence of Alterations in Fluorescent In Situ Hybridisation (FISH) of Spermatozoa and to Evaluate the Efficacy of the Use of Annexin Columns (MACS®) in Patients With Altered FISH Undergoing In Vitro Fertilisation Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria y Biomédica de Alicante (Network)
Responsible Party: Principal Investigator, Borja Tejero Llinares, Biologist, Instituto de Investigación Sanitaria y Biomédica de Alicante
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 190767
Record Dates: First submitted 2024-07-21; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Infertility, Male
Keywords: In Vitro Fertilization; sperm FISH; annexin columns; MACS; Preimplantation Genetic Testing for aneuploidies
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Intervention Model Description: A total of 10 couples with no previous children in common, negative serology and normal karyotype were included. Females were aged less than 40 years and males less than 50 years at the time of treatment.
  The semen sample of each couple was capacitated by density gradient centrifugation (DGC) and swim up, forming the control group. An aliquot was taken that was destined to pass through the annexin columns (MACS® ART, Miltenyl Biotic GmbH, Germany) constituting the study group. The oocytes obtained in each of the couples were pseudo-randomized and inseminated by ICSI with sperm from the study group and the control group. All couples benefited from the experimental treatment since they had the opportunity to inseminate their oocytes with sperm from both groups, thus excluding treatment bias or asymmetry.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Access to the data was restricted to the study investigators, health authorities and ISABIAL advisory bodies, when necessary, to check the study data and procedures, but always maintaining confidentiality.
  The data collected for the study was identified by a code, so that no information that could identify the participants was included, and only the researchers were able to link the anonymized data to the clinical history.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MACS (Experimental): Oocytes corresponding to this group were inseminated by spermatozoa selected after the use of MACS.
  Interventions: Device: Magnetic Activated Cell Sorting
- Control (No Intervention): Oocytes corresponding to this group were inseminated with spermatozoa obtained after density gradient centrifugation.

INTERVENTIONS:
Device: Magnetic Activated Cell Sorting — The MACS® ART Annexin V System has been designed for the in vitro elimination of apoptotic human spermatozoa in fresh, cryopreserved or otherwise manipulated semen samples. Samples processed by this technique can be subsequently used in any assisted reproduction procedure.
  Annexin V recognizes externalized phosphatidylserine (ePS) on the plasma membrane of apoptotic spermatozoa. Depletion of the altered sperm begins with magnetic tagging of the sperm. The system selectively retains unwanted sperm by utilizing the natural ability of annexin V to recognize the ePS on the plasma membrane of the altered sperm, because annexin V is conjugated to metal microspheres. The labeled cells pass through a separation column in a fixed magnetic field. Unwanted (altered) spermatozoa are selectively retained in the separation column. Unlabeled spermatozoa pass through the column where they are collected for later use.
  Other Names: MACS
  Arms: MACS

SUMMARY:
250 petitions for FISH of spermatozoa were requested, determining the total and particular incidence in each of the indications collected. The effect of annexin columns was evaluated in 10 couples with altered FISH. In each of the couples, oocytes were pseudo-randomised to the control group and MACS®. All couples received experimental treatment. Mixed logistic regression model were adjusted to evaluate the effect of MACS® on the response variables studied.

DETAILED DESCRIPTION:
Prospective pseudo-randomised study carried out in the reproduction unit of the Hospital General Universitario Dr. Balmis in Alicante. The study was divided into two phases, with both being conducted in parallel. The research was approved by the Ethics Committee for Research on Medicines (CEIm) of the Alicante Department of Health. The treatment and use of the clinical data required for this study complied with current legislation, preserving the anonymity of the patients.

Phase I. A total of 250 sperm FISH tests were requested for different indications in men aged 18-55 years with normal karyotype. Of the total number of tests requested, 16 could not be performed due to low sperm count. Finally, 234 samples were analysed, of which 20 had altered sperm FISH.

Phase II. From the previous phase, not all patients with an altered FISH test were included in the second phase of the study, some of them were lost for different reasons (n=10). A total of 10 couples with no previous children in common, negative serology and normal karyotype were included. Females were aged less than 40 years and males less than 50 years at the time of treatment.

The semen sample of each couple was capacitated by density gradient centrifugation (DGC) and swim up, forming the control group. An aliquot was taken that was destined to pass through the annexin columns (MACS® ART, Miltenyl Biotic GmbH, Germany) constituting the study group. The oocytes obtained in each of the couples were pseudo-randomized and inseminated by ICSI with sperm from the study group and the control group. All couples benefited from the experimental treatment since they had the opportunity to inseminate their oocytes with sperm from both groups, thus excluding treatment bias or asymmetry.

To evaluate the efficacy of MACS® on laboratory outcome, fertilization rates, abnormal fertilization, biopsiable embryos and euploid embryos were compared between the study and control group.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 40 years of age. Men between 18 and 55 years of age.
* Couples without any common, previous and healthy children.
* Couples with indication of IVF-ICSI cycle with Preimplantation Genetic Test for Aneuploidy (PGT-A).
* Men with altered sperm FISH results.

Exclusion Criteria:

* Prior voluntary sterilization.
* Existence of documented medical contraindication for infertility treatment.
* Existence of documented medical contraindication to pregnancy.
* Existence of a documented medical situation that seriously interferes with the development of the offspring.
* Impossibility to comply with the treatment for health-related reasons or other family or social environment-related reasons.
* Existence of a documented situation referring to any other circumstance that may seriously interfere with the development of the offspring submitted for consideration to a health care ethics committee or similar body.
* One or both partners with positive serology for HIV, HBV and VDRL.
* One or both partners with partner with altered karyotype.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Euploid embryo rate | This variable was taken 2 days after obtaining the genetic result of the embryo biopsy.
  Embryos without chromosomal alterations in relation to the total number of those that were informative.

SECONDARY OUTCOMES:
Fertilization rate | This variable was taken 17-20 hours after oocyte insemination.
  Number of correctly fertilized zygotes among the total number of mature oocytes inseminated
Biopsiable embryo rate | This variable was taken on the 3rd day of embryonic development, at the time of the embryo biopsy. .
  Number of biopsied embryos versus the total number of correctly fertilized zygotes

CONTACTS AND LOCATIONS:
Locations (1):
- ISABIAL, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No